CLINICAL TRIAL: NCT05924607
Title: Comparative Effects of Clamshells Exercise and Vastrus Medialis Oblique Strengthening Exercise on Patellofemoral Pain Syndrome
Brief Title: Clamshells Exercise and Vastrus Medialis Oblique Strengthening Exercise on Patellofemoral Pain Syndrome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR & AHS/23/0101
Record Dates: First submitted 2023-04-18; First posted 2023-06-29 (Actual); Last update posted 2023-06-29 (Actual); Status verified 2023-06

CONDITIONS: Patellofemoral Pain Syndrome
MeSH Terms: conditions — Patellofemoral Pain Syndrome

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard clamshells method (Experimental): The patient is asked to lie in a side-lying position with the weak limb up, both hips flexed at 45°, the knees flexed at 90°, and neither the feet nor back not in contact with the wall. Keeping both their heels and the first metatarsal head together, the patient separated their knees and rotated the weak limb upward. The patients is instructed not to tip it backward and to hold the pelvis in a neutral position.Common treatment will be given to each patient includes hot pack for 10 minutes and knee isometric contraction exercises and SLR( 3-5 sets of 10 repetitions)
  Interventions: Other: Standard clamshells method
- Targeted VMO strengthening (Experimental): The patient is asked to lie in a supine lying position with arm next to the body. After that asked the patient to perform SLR exercise in an external hip rotation with the simultaneous contraction of the ankle dorsiflexors. Common treatment will be given to each patient includes hot pack for 10 minutes and knee isometric contraction exercises and SLR( 3-5 sets of 10 repetitions
  Interventions: Other: Targeted VMO strengthening

INTERVENTIONS:
Other: Standard clamshells method — The patient is asked to lie in a side-lying position with the weak limb up, both hips flexed at 45°, the knees flexed at 90°, and neither the feet nor back not in contact with the wall. Keeping both their heels and the first metatarsal head together, the patient separated their knees and rotated the weak limb upward. The patients is instructed not to tip it backward and to hold the pelvis in a neutral position
  Arms: Standard clamshells method
Other: Targeted VMO strengthening — Targeted VMO strengthening The patient is asked to lie in a supine lying position with arm next to the body. After that asked the patient to perform SLR exercise in an external hip rotation with the simultaneous contraction of the ankle dorsiflexors. Common treatment will be given to each patient includes hot pack for 10 minutes and knee isometric contraction exercises and SLR( 3-5 sets of 10 repetitions
  Arms: Targeted VMO strengthening

SUMMARY:
PFPS, also known as patellofemoral pain syndrome, is a prevalent musculoskeletal condition that primarily affects adolescents and young adults. When engaging in various activities, such as stair climbing, running, jumping, kneeling, or prolonged sitting, it is characterized by aching pain in the peripatellar region. Any disruption of these would result in abnormal PFJ overloading. Normal patellar tracking on the trochlea groove relies on the coordination and balance of many structures, including soft tissues, muscles, tendons, ligaments, and the shape of articular surfaces around the knee joint. Research in a variety of fields has received support the therapeutic exercise known as "clamshells" for stabilizing the pelvis by strengthening the hip abductors and external rotators.VMO strengthening exercises are also essential in keeping the patella in the trochlear groove and lowering the lateral vector force on the patellofemoral joint. This research aims to evaluate the effects of clamshells exercise and Vastrus medialis oblique strengthening exercise in patients with Patellofemoral pain syndrome.

The study would be randomized clinical trial. Total fourty two subjects will be assigned randomly by using lottery method into two groups. Group A will be given clamshell exercise with baseline treatment while Group B will receive targeted vastrus medialis oblique strengthening exercise with baseline treatment. After confirmation of diagnosis with physical examination as well as zohlar's test /20 cm step down test are recommended. Numeric pain rating scale (NPRS) and Lower extremity functional scale (LEFS) would be used as an outcome measure tools for pain and functional limitation respectively. Measurements will be taken at (Baseline and at the end of treatment session). The collected data will be analyzed in Statistical Package for the Social Sciences (SPSS) 25.0. Parametric/non-parametric tests will be applied after testing normality of data.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 40years
* Both Genders (male & female)
* Unilateral or bilateral knee pain for at least 1-3 month,
* Pain provoked by at least 3 functional activities ( ascending/descending stairs, kneeling, jumping, running, squatting,hopping,prolonged sitting)
* Average NPRS score above 3 out of 10 during previous week.
* Knee pain on stepping down from 20cm step height.

Exclusion Criteria

* Previous history of patellar subluxation or dislocation
* Knee surgery within previous year
* History of knee joint pathologies ( meniscus,ligament injuries,)
* Any fracture of lower extremity
* Massive effusion/any abnormal deformity of knee joint.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 42 (Estimated)
Dates: Start 2022-11-14 (Actual); Primary Completion 2023-08-24 (Estimated); Study Completion 2023-08-30 (Estimated)

PRIMARY OUTCOMES:
Pain intensity | Baseline to 6th week
  numeric pain rating scale(NPRS) is used to measure intensity of pain.Score ranges from 0-10.Higher values mean greater level o pain.
Functional disability | Baseline to 6th week
  The lower Extremity Functional Scale (LEFS) is used to measure the functional status of the lower extremity. score ranges from 0-80. lower values mean greater functional limitation.
Muscle strength | Baseline to 6th week
  Sphygmomanometer is used to measure muscle strength. higher readings on sphygmomanometer represents better muscle strength.

CONTACTS AND LOCATIONS:
Overall Officials: Dr.Rabiya Noor, Phd, Principal Investigator — Riphah International University
Locations (1):
- Ittefaq Hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hott A, Brox JI, Pripp AH, Juel NG, Liavaag S. Patellofemoral pain: One year results of a randomized trial comparing hip exercise, knee exercise, or free activity. Scand J Med Sci Sports. 2020 Apr;30(4):741-753. doi: 10.1111/sms.13613. Epub 2020 Jan 5. PMID 31846113
- [Background] Foroughi F, Sobhani S, Yoosefinejad AK, Motealleh A. Added Value of Isolated Core Postural Control Training on Knee Pain and Function in Women With Patellofemoral Pain Syndrome: A Randomized Controlled Trial. Arch Phys Med Rehabil. 2019 Feb;100(2):220-229. doi: 10.1016/j.apmr.2018.08.180. Epub 2018 Sep 26. PMID 30267667
- [Background] Azab AR, Abdelbasset WK, Basha MA, Mahmoud WS, Elsayed AE, Saleh AK, Elnaggar RK. Incorporation of Pilates-based core strengthening exercises into the rehabilitation protocol for adolescents with patellofemoral pain syndrome: a randomized clinical trial. Eur Rev Med Pharmacol Sci. 2022 Feb;26(4):1091-1100. doi: 10.26355/eurrev_202202_28098. PMID 35253163